CLINICAL TRIAL: NCT01563536
Title: An Open-Label, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of ABT-267 in HCV Infected Subjects
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of ABT-267 in HCV Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-386
Record Dates: First submitted 2012-01-27; First posted 2012-03-27 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2014-12

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C,Genotype 1
MeSH Terms: interventions — ombitasvir; paritaprevir; dasabuvir; Ritonavir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABT-267 1.5 mg, then ABT-267, ABT-450/r, ABT-333, plus RBV (Experimental): ABT-267 (1.5 mg once daily) as monotherapy for 2 days, then ABT-267 (1.5 mg once daily), ABT-450/r (150 mg/ 100 mg once daily) and ABT-333 (400 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) combination therapy for 12 weeks
  Interventions: Drug: ABT-267; Drug: ABT-450; Drug: ABT-333; Drug: Ritonavir; Drug: Ribavirin
- ABT-267 25 mg, then ABT-267, ABT-450/r, ABT-333, plus RBV (Experimental): ABT-267 (25 mg once daily) as monotherapy for 2 days, then ABT-267 (25 mg once daily), ABT-450/r (150 mg/ 100 mg once daily) and ABT-333 (400 mg twice daily), plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) combination therapy for 12 weeks
  Interventions: Drug: ABT-267; Drug: ABT-450; Drug: ABT-333; Drug: Ritonavir; Drug: Ribavirin

INTERVENTIONS:
Drug: ABT-267 — Tablet
  Other Names: ombitasvir
Drug: ABT-450 — Tablet
Drug: ABT-333 — Tablet
  Other Names: dasabuvir
Drug: Ritonavir — Capsule
Drug: Ribavirin — Tablet

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, and antiviral activity of multiple, ascending doses of ABT-267 (also known as ombitasvir) administered as two-day monotherapy followed by ABT-267 in combination therapy with other direct-acting antiviral agents (DAAs) ABT-450 with ritonavir (ABT-450/r) and ABT-333 (also known as dasabuvir) plus ribavirin (RBV) in patients with chronic Hepatitis C virus (HCV) infection without cirrhosis.

DETAILED DESCRIPTION:
An open-label, multicenter study to evaluate the safety, tolerability, pharmacokinetics, and antiviral activity of ABT-267 as monotherapy for 2 days, followed by ABT-267, ABT-450 with ritonavir (ABT-450/r) and ABT-333 plus ribavirin (RBV) combination therapy for 12 weeks in treatment-naïve, non-cirrhotic patients with chronic hepatitis C virus (HCV) infection. The study included post-treatment follow-up for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age of 18 and 70 years, inclusive, at time of enrollment.
* Subject has never received antiviral treatment for hepatitis C virus (HCV) infection.
* Body mass index (BMI) is ≥ 18 to < 38 kg/m^2. BMI is calculated as weight measured in kilograms (kg) divided by the square of height measured in meters (m).
* Chronic HCV genotype 1-infection for at least 6 months prior to study enrollment.
* Subject has plasma HCV RNA level > 10,000 IU/mL at screening

Exclusion Criteria:

* History of severe, life-threatening or other significant sensitivity to any drug.
* Females who are or plan to become pregnant or breastfeeding or males whose partner is pregnant or planning to become pregnant.
* Recent history of drug or alcohol abuse that could preclude adherence to the protocol.
* Positive test result for hepatitis B surface antigen or anti-human immunodeficiency virus (HIV) antibodies.
* Any current or past clinical evidence of cirrhosis (e.g., ascites, esophageal varices), or a liver biopsy or FibroTest/aspartate aminotransferase to platelet ratio (APRI) or FibroScan® showing cirrhosis or extensive bridging fibrosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L Campbell, MD, Study Director — AbbVie
Locations (4):
- United States (4):
  - Site Reference ID/Investigator# 68002, Bakersfield, California
  - Site Reference ID/Investigator# 67383, Orlando, Florida
  - Site Reference ID/Investigator# 67382, Annapolis, Maryland
  - Site Reference ID/Investigator# 67385, Poughkeepsie, New York

REFERENCES:
- [Background] Mensing S, Polepally AR, Konig D, Khatri A, Liu W, Podsadecki TJ, Awni WM, Menon RM, Dutta S. Population Pharmacokinetics of Paritaprevir, Ombitasvir, Dasabuvir, Ritonavir, and Ribavirin in Patients with Hepatitis C Virus Genotype 1 Infection: Combined Analysis from 9 Phase 1b/2 Studies. AAPS J. 2016 Jan;18(1):270-80. doi: 10.1208/s12248-015-9846-1. Epub 2015 Nov 23. PMID 26597291
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Started | 6 | 6
Completed | 5 | 4
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (4.76) | 46.8 (11.84) | 49.2 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of ABT-267 Following Monotherapy on Day 1
Description: Blood samples were collected pre-dose (time 0) and at 2, 4, and 6 hours post-dose on Day 1 and pre-dose on Day 2 (ABT-267 monotherapy). The samples were analyzed for ABT-267 using validated analytical methods. Maximum plasma concentration (Cmax; measured in ng/mL) was estimated using noncompartmental analyses.
Time Frame: Day 1 (pre-dose [time 0] and at 2, 4, and 6 hours post-dose) and Day 2 (pre-dose)
Population: All participants who received at least one dose of study drug (intent-to-treat [ITT] population).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
ng/mL | 1.66 (0.21) | 41.0 (16.5)

2. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of ABT-267 Following Monotherapy on Day 1
Description: Blood samples were collected pre-dose (time 0) and at 2, 4, and 6 hours post-dose on Day 1 and pre-dose on Day 2 (ABT-267 monotherapy). The samples were analyzed for ABT-267 using validated analytical methods. Time of maximum plasma concentration (Tmax; measured in hours) was estimated using noncompartmental analyses.
Time Frame: Day 1 (pre-dose [time 0] and at 2, 4, and 6 hours post-dose) and Day 2 (pre-dose)
Population: All participants who received at least one dose of study drug (ITT population).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
hours | 3.67 (0.82) | 3.67 (1.5)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours (AUC[24]) of ABT-267 Following Monotherapy on Day 1
Description: Blood samples were collected pre-dose (time 0) and at 2, 4, and 6 hours post-dose on Day 1 and pre-dose on Day 2 (ABT-267 monotherapy). The samples were analyzed for ABT-267 using validated analytical methods. Area under the plasma concentration-time curve from time 0 to 24 hours (AUC[24]; measured in ng multiplied by hour/mL) was estimated using noncompartmental analyses.
Time Frame: Day 1 (pre-dose [time 0] and at 2, 4, and 6 hours post-dose) and Day 2 (pre-dose)
Population: All participants who received at least one dose of study drug (ITT population).
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 18.0 (2.46) | 467 (236)

4. Primary Outcome: Plasma Concentration of ABT-267 Pre-dose (Ctrough) on Day 2 and Day 3
Description: Blood samples were collected pre-dose on Day 2 (prior to second dose of ABT-267 monotherapy) and pre-dose on Day 3 (prior to first dose of combination therapy). The samples were analyzed for ABT-267 using validated analytical methods. Pre-dose plasma concentrations on Day 2 and Day 3 (Ctrough, measured in ng/mL) are reported.
Time Frame: Day 2 (pre-dose) and Day 3 (pre-dose)
Population: All participants who received at least one dose of study drug (ITT population).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 2 Ctrough | 0 (0) | 5.2 (1.78)
  Day 3 Ctrough | 0.228 (0.263) | 6.62 (3.77)

5. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this treatment.
  The investigator assessed the relationship of each AE to the use of direct-acting antiviral agents (DAAs), and rated the severity of each event as either: Mild: The AE was transient and easily tolerated by the participant; Moderate: The AE caused the participant discomfort and interrupted usual activities; Severe: The AE caused considerable interference with the participant's usual activities and could have been incapacitating or life-threatening.
  A serious adverse event was any event that resulted in death, was life-threatening, resulted in hospitalization or prolongation of hospitalization, resulted in a congenital anomaly or persistent or significant disability or was any other important medical event requiring medical or surgical intervention.
Time Frame: All AEs were collected from the time of study drug administration to 30 days after last dose of study drug (16 weeks).
Population: All participants who received at least one dose of study drug (safety population).
Measure: Number; unit: participants
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
participants
  Any AE | 3 | 5
  Any AE at least possibly related to DAAs | 3 | 4
  Any severe AE | 0 | 1
  Any serious AE | 0 | 2
  Any AE leading to discontinuation of study drug | 0 | 1
  Any AE leading to interruption of study drug | 0 | 0
  Any AE leading to RBV dose modification | 0 | 1
  Any fatal AE | 0 | 0
  Deaths | 0 | 0

6. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks and 24 Weeks After Combination Therapy
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 12 and 24 weeks after the last dose of combination study drug. The LLOQ for the assay was 25 IU/mL.
Time Frame: 12 and 24 weeks after last dose of combination study drug
Population: All participants who received at least one dose of study drug (ITT population); participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
percentage of participants
  12 Weeks Post-treatment | 83.3 | 83.3
  24 Weeks Post-treatment | 83.3 | 83.3

7. Secondary Outcome: Percentage of Participants With Rapid Virologic Response
Description: The percentage of participants with virologic response (plasma HCV RNA less than the lower limit of quantitation [< LLOQ]) after 4 weeks of combination therapy.
Time Frame: 4 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
percentage of participants | 83.3 | 100

8. Secondary Outcome: Percentage of Participants With End-of-Treatment Response
Description: The percentage of participants with virologic response (plasma HCV RNA less than the lower limit of quantitation [< LLOQ]) at the end of combination therapy (12 weeks).
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
percentage of participants | 83.3 | 83.3

9. Secondary Outcome: Percentage of Participants With Extended Rapid Virologic Response
Description: The percentage of participants with virologic response (plasma HCV RNA less than the lower limit of quantitation [< LLOQ]) at Weeks 4 through 12 of combination therapy.
Time Frame: Weeks 4 to 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
percentage of participants | 83.3 | 83.3

10. Secondary Outcome: Mean Change in Viral Load From Baseline to Pre-dose on Day 2 and Day 3 of ABT-267 Monotherapy
Description: The relationship between ABT-267 dose, ABT-267 concentration, and response was analyzed as the change in viral load (measured as log10 IU/mL) from baseline (pre-dose on Day 1) to pre-dose on Days 2 and 3. Plasma concentrations of ABT-267 pre-dose on Days 2 and 3 are presented above in 4. Primary Outcome: Plasma Concentration of ABT-267 Pre-dose (Ctrough) on Day 2 and Day 3.
Time Frame: Predose on Days 1, 2, and 3
Population: All participants who received at least one dose of study drug (ITT population).
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
log10 IU/mL
  Day 2 Mean change in Viral Load from Baseline | -1.95 (0.630) | -2.85 (0.421)
  Day 3 Mean change in Viral Load from Baseline | -1.96 (0.405) | -3.10 (0.257)

11. Primary Outcome: Mean Maximal Decrease From Baseline in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) During ABT-267 Monotherapy
Description: The baseline value was the last measurement before the first dose of ABT-267 monotherapy (Day 1). The maximal decrease during monotherapy was the change from baseline to the lowest log10 IU/mL HCV RNA level any time from the first dose of ABT-267 on Day 1 to the last log10 HCV RNA level before the first dose of ABT-267 combination therapy (Study Day 3).
Time Frame: Pre-dose on Days 1, 2, and 3
Population: All participants who received at least one dose of study drug (ITT population).
Measure: Least Squares Mean (Standard Error); unit: log10 IU/mL
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
log10 IU/mL | -1.6 (0.41) | -3.1 (0.41)
Statistical Analysis 1: Comparison: ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV vs ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV; Test type: Superiority or Other; p = 0.035, ANCOVA — Pre-specified 2-sided significance level of 0.05; Analysis of covariance (ANCOVA) with the baseline log10 HCV RNA values as a covariate and with an effect for treatment arm; Mean Difference (Maximal Decrease) = -1.5, 95% CI 2-sided [-2.81 to -0.13]

12. Other Pre Specified Outcome: Resistance-Associated Variants and Phenotypic Resistance
Description: Baseline (pre-dose on Day 1) samples were analyzed for resistance-associated amino acid (AA) variants using population sequencing. Phenotypic resistance to ABT-267 at Baseline was assessed by calculating the fold difference in the the half maximal effective concentration (EC50) compared with the EC50 for the appropriate reference replicon (1a-H77 or 1b-Con1). Day 3 samples were analyzed using population sequencing and were compared with the baseline and appropriate prototypic reference sequences to assess AA changes. Phenotypic resistance at Day 3 was assessed by calculating the fold difference in the EC50 compared with the EC50 for the corresponding Baseline sample. The number of participants with variants at resistance-associated AA positions and phenotypic resistance at Baseline and Day 3 are presented.
Time Frame: Day 1 Pre-dose (Baseline) and Day 3 Pre-dose
Population: All participants who received at least one dose of study drug (ITT population) and had evaluable data were analyzed for baseline resistance-associated amino acid variants; the development of viral resistance was analyzed in all participants who received at least 1 dose of ABT-267 whose samples had sufficient viral titer to allow analysis.
Measure: Number; unit: participants
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Number analyzed (Participants) | 6 | 6
participants
  Baseline Variants in NS5A (n=5, 6) | 2 | 0
  Baseline Resistance >10-fold (n=5, 6) | 1 | 0
  Day 3 Variants in NS5A (n=5, 2) | 6 | 2
  Day 3 Resistance >10-fold (n=5, 2) | 1 | 2

ADVERSE EVENTS:
Time Frame: All AEs were collected from the time of study drug administration to 30 days after last dose of study drug (16 weeks); SAEs were also collected from the time that informed consent was obtained until the end of the study (60 weeks).
Arm/Group | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/6
Other Adverse Events (participants affected / at risk) | 3/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV (N=6) | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV (N=6)
LABYRINTHITIS (Infections and infestations) | 0 | 1
MANIA (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-267 1.5 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV (N=6) | ABT-267 25 mg, Then ABT-267, ABT-450/r, ABT-333, Plus RBV (N=6)
TACHYCARDIA (Cardiac disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 2
DRY MOUTH (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1
ASTHENIA (General disorders) | 0 | 1
CHEST PAIN (General disorders) | 0 | 1
FATIGUE (General disorders) | 1 | 2
GASTROENTERITIS (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 2
HAEMOGLOBIN DECREASED (Investigations) | 0 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
BURNING SENSATION (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 2
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 | 0
ABNORMAL DREAMS (Psychiatric disorders) | 1 | 1
SLEEP DISORDER (Psychiatric disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.